CLINICAL TRIAL: NCT05560256
Title: Building Capacity in Human-Centered Design: Developing a Diabetes Mobile Health Application for and With Kenyan Adolescents
Brief Title: Developing a Diabetes Mobile Health Application for and With Kenyan Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Kenyan Diabetes Management & Information Centre (DMI) (Unknown)
Responsible Party: Principal Investigator, Susan Wyche, Associate Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1R21TW011339-01 (NIH)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes
Keywords: Human-Centered Design; Mobile Phones; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Masking Description: We asked participants to interact with the paper diary during a workshop.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth Engage with Diary (Experimental): 24 youth will use the Diary for one month
  Interventions: Other: Diary/Journal

INTERVENTIONS:
Other: Diary/Journal — Participants will be given a diary to record their blood glucose measurements, and other pertinent information (diet and activities).
  Other Names: Diary

SUMMARY:
With over 6 billion mobile phone subscribers and 75% of the world having access to a device, global health communities increasingly recognize the potential for using these devices to improve access to health care and health outcomes-especially in sub-Saharan Africa (SSA), where device ownership has grown dramatically. Less attention, however, has been given to developing the research capacity to allow these countries' public health researchers to collaborate with software developers and the users of mobile health applications (henceforth apps) to develop their own interventions. If mobile health apps are to be adopted, effective, and scalable, they must be designed by and with these individuals, the people most knowledgeable about the issues affecting technology use and disease management in their countries. Human-centered design (HCD), or design thinking, is a promising design strategy that prioritizes the needs of the intended population. It has also been successfully used to develop innovative and locally relevant health interventions that improve health outcomes. The purpose of this R21 proposal is to introduce Kenyan public health researchers and software developers to the HCD process and then collaboratively develop and evaluate an mobile health app that targets a growing epidemic among middle-to-late adolescents (13-18 yrs.) in Kenya-Type 1 Diabetes (T1D). To achieve this goal, we will pursue these specific aims: (1) train Kenyan health practitioners and software developers in HCD; (2) use HCD to build a prototype mHealth intervention for adolescents in Kenya with T1D; and (3) assess the prototype's usability, accessibility, and feasibility in using it to increase adolescents' knowledge of T1D and management of the disease. Our long-term goals include: (1) building research capacity by establishing a research network between health researchers at The Kenyan Diabetes Management and Information Center (DMI-a non-profit organization that works with adolescents with T1D) and mobile software developers at Lake Hub (an innovation space) so they can design future mobile health apps; (2) developing a commercially available app that Kenyan adolescents can use to manage T1D and stay healthy; and (3) evaluating the HCD process as it applies to developing mobile health interventions that improve health outcomes.

DETAILED DESCRIPTION:
Aim #1 Train Kenyan health practitioners and software developers in HCD. We accomplished this by implementing an HCD curriculum during a three-day workshop with our Kenyan collaborators. Drs. Wyche, Olson and Holtz, travelled to Nairobi, Kenya, between September 28 and October 5 to conduct our three-day training workshop. Our collaborators from LakeHub (in Kisumu) also flew to Nairobi. Our other collaborators-from DMI-are based in Kenya's capital city. We held the workshop at the Ngong Hills Hotel in Nairobi.

Aim #2 Use HCD to build a prototype intervention for adolescents in Kenya with T1D. We accomplished this aim by conducting interviews; analyzing data; holding two design workshops; developing an initial version of a diary; conducting a pilot evaluation of the diary; and iterating upon the diary's design. Significant project outcomes include a personal diary.

In April 2022, Dr. Jennifer Olson, and our collaborators at DMI and ROA, interviewed 24 youth with T1D at two sites in Kenya (Vihiga County and Nairobi); 12 participants in each site. She also interviewed their parents/caregivers (n=22), as well as key stakeholders (e.g., doctors, teachers, community health workers). Interviews were digitally recorded (with participants' consent). During this time, we also provided youth with a digital camera and asked them to engage in a photovoice exercise (i.e., asking participants to take photographs, and then reflecting upon the reasons, emotions and experiences that motivated them to take the photos).

We hired translators-fluent in Kiswahili and English-to translate and transcribe the interviews. We also collected participants' photographs. Drs. Olson and Wyche analyzed this transcribed interviews and photographs in May-June 2022. Our objective was to deepen our understanding of how youth managed T1D and to identify possible technology interventions. A significant finding was that developing a mobile phone application would not support youths' existing practices. Most participants are not allowed to use mobile phones in school. Further, not all participants, especially those living in rural areas, had access to a smart phone.

In July 2022, Drs. Wyche and Olson travelled to Kenya. We held two, two-day design workshops (between July 3 and July 7). The first was held at Sosa Cottages (Majengo); the second was held at Ngong Hills Hotel (Nairobi). All of the youth and caregivers, who Dr. Olson interviewed in April, attended the workshops. Workshop objectives included: learning more about youth and T1D; and brainstorming design interventions that would help youth manage the disease. During these sessions, participants discussed their experiences managing T1D; they also talked about their photographs. Other significant activities include brainstorming exercises. Participants ideas included posters that would educate people about T1D, a calendar that would help youth keep track of their doctors' appointments, and diary that supported T1D-related activities. At the conclusion of the workshops Drs. Wyche and Olson determined that the diary was the most promising intervention. The diary would allow youth to track their sugar levels, as well as what they ate and their activity levels. The diary would also include useful information about how to effectively manage T1D (e.g., how to inject insulin, to make healthy meals, and properly store insulin). They worked with designed from LakeHub to develop an initial version of this diary.

In September 2022, the design team printed 60 initial copies of the diary. During this time, Drs. Wyche and Olson returned to Kenya to share these diaries with doctors, our collaborators (at DMI and ROA), and with the youth and their caregivers. Dr. Wyche met with Drs. Karakezi and Ngugi (DMI) to review the text in the diary. We also held two, daylong workshops-one in Vihiga and one in Nairobi-to introduce the diary to the youth and their parents. Our objective was to get preliminary feedback on how to improve the diary's design. Outcomes of these interviews and workshops included significant insights about changes that would improve the diary (e.g., modifying text, changing images, adding more information).

Aim #3 The final phase of the HCD process is implementation, or the project's formative evaluation phase. In September 2022, we gave the prototype diary to the youth, their caregivers, and other stakeholders who contributed to its development (e.g., doctors, and community health workers). Our objective was to validate the intervention's usefulness as well as the feasibility of using it to increase adolescents' knowledge of T1D and management of the disease. To achieve this goal, we conducted focus groups to assess youth's initial reactions to the diary, asked them to fill out pages (e.g., blood glucose monitoring page), and solicited feedback on the diary's strengths and weaknesses. We also administered a short survey to assess how often the diary was used during a one-month period. Participants' feedback was generally positive. They commented on the diary's professional appearance and noted the inclusion of images that were similar to their context (e.g., illustrations of foods they ate). We also received significant feedback on how to improve the diary. This included adding more information about how to properly store insulin-when you do not have access to a refrigerator-as well as guidance on how to best inject insulin. Survey data suggested frequent use of the diary (i.e., at least once a day).

ELIGIBILITY:
Inclusion Criteria:

* T1D diagnosis 13-18 years old
* Have an A1c > 7
* Uses a phone
* Fluent in Swahili

Exclusion Criteria:

* Being treated for significant medical condition other than T1D
* Being treated for eating disorder

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Building Capacity in Human-Centered Design: Developing a Diabetes mHealth Application for and with Kenyan Adolescents | 1 month
  Feasibility of Diary

CONTACTS AND LOCATIONS:
Locations (1):
- Nairobi, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No